CLINICAL TRIAL: NCT04136704
Title: Long-Term Outcomes of Sleeve Gastrectomy in Children and Adolescents
Brief Title: Long-Term Outcomes of LSG in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Collaborators: New You Medical Center (Unknown)
Responsible Party: Principal Investigator, Aayed Alqahtani, Professor of Surgery, King Saud University
Other Study IDs: LSGKids10
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Obesity, Childhood; Bariatric Surgery Candidate; Cardiovascular Risk Factor
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, subcutaneous and visceral fat, and liver samples obtained from patients who consent to have sample storage in liquid nitrogen for research purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Sleeve Gastrectomy in Pediatric Patients: Laparoscopic Sleeve Gastrectomy will be offered as an adjuvant to a multidisciplinary family-based program that focuses on nutrition, physical activity, and behavioral counseling.
  Interventions: Procedure: Sleeve gastrectomy
- Sleeve Gastrectomy in Adult Patients: This comparison group will be composed of adult patients who undergo sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic sleeve gastrectomy
  Other Names: Vertical Sleeve Gastrectomy

SUMMARY:
This project aims to assess the short- and long-term safety and efficacy of bariatric surgery in children and adolescents compared to adults.

DETAILED DESCRIPTION:
Obesity affects children and adults across all age groups. More than 30% of children and adolescents in the United States are currently overweight or obese, whereas the prevalence of obesity is as high as 21.4% in young children.This increase in prevalence is associated with significant short- and long-term health implications and necessitates effective interventions that induce significant weight loss and ameliorate associated conditions.

The results of weight loss surgery in children and adolescents are still scarce, despite recent studies suggesting favorable short- and intermediate-term outcomes that are comparable to those in adults. Although evidence continues to emerge, this solution is still denied to young children.

Bariatric surgery has proven safety and efficacy in inducing significant weight loss and co-morbidity resolution in children and adolescents. However, long-term evidence in this age group is yet to be reported. This project aims to study long-term weight loss, cardiovascular risk factors, growth and morbidity in severely obese children and adolescents (aged 5-21 years) who undergo laparoscopic sleeve gastrectomy (LSG).

This study aims to narrow the current evidence gap by studying the long-term effects of bariatric surgery in children and adolescents with severe obesity.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 5 to 21 years
* BMI higher than the 140% of the 95th percentile for age and gender
* failure to lose satisfactory weight during a period of at least 6 months
* Supportive psychological evaluation
* Presence of a dedicated caretaker from the patient's family
* Motivation, realistic expectations
* Informed consent or assent with concomitant parental consent for patients aged < 17 years
* Absence of medical and surgical contraindications

Exclusion Criteria:

* Cardiac failure
* Respiratory failure
* Immune deficiency
* GI disease
* Age greater than 21 years
* Inability to sign informed consent / assent

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents who meet the inclusion criteria, fail to lose weight under an intensive family-based nutrition and lifestyle program, who signed an informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Weight Change | Calculated at each follow-up milestone up to 10 years
  Weight change according to %excess weight loss (%EWL), %BMI change, % total weight loss (%TWL), BMI change, BMI z-score change
Growth | Calculated at each follow-up milestone up to 10 years
  Measurement of change in growth velocity (height z-score change)
Remission of Type 2 Diabetes | Predetermined follow-up intervals up to 10 years, i.e. short-term: 1-3 years; medium-term: 4-6 years; long-term: 7-10 years
  Remission of type 2 diabetes is assessed in accordance with the American Society for Metabolic and Bariatric Surgery (ASMBS) Outcomes Reporting Standards
% Change in Framingham 30-Year Cardiovascular Disease (CVD) Risk | Predetermined follow-up intervals up to 10 years, i.e. short-term: 1-3 years; medium-term: 4-6 years; long-term: 7-10 years
  Proportion of patients at risk for a full CVD event according to the Framingham 30-year risk score for CVD at baseline and follow-up
Proportion of participants reporting adverse events | 30-day morbidity and mortality, and events reported during predetermined follow-up intervals up to 10 years, i.e. short-term: 1-3 years; medium-term: 4-6 years; long-term: 7-10 years
  Number of participants with grade 2 or higher complication according to Clavien-Dindo Classification
Number of participants undergoing a reoperative or revisional surgical or endoscopic intervention | Predetermined follow-up intervals up to 10 years, i.e. short-term: 1-3 years; medium-term: 4-6 years; long-term: 7-10 years
  Number of participants who underwent reoperation, defined as undergoing subsequent abdominal surgery for sleeve gastrectomy related complications, and revision, defined as undergoing a subsequent bariatric or endobariatric procedure to re-induce weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Aayed R Alqahtani, MD, Study Chair — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elahmedi MO, Alqahtani AR. Evidence Base for Multidisciplinary Care of Pediatric/Adolescent Bariatric Surgery Patients. Curr Obes Rep. 2017 Sep;6(3):266-277. doi: 10.1007/s13679-017-0278-3. PMID 28755177
- [Background] Alqahtani AR, Elahmedi M, Alqahtani YA. Bariatric surgery in monogenic and syndromic forms of obesity. Semin Pediatr Surg. 2014 Feb;23(1):37-42. doi: 10.1053/j.sempedsurg.2013.10.013. Epub 2013 Nov 15. PMID 24491367
- [Result] Alqahtani A, Elahmedi M, Alswat K, Arafah M, Fagih M, Lee J. Features of nonalcoholic steatohepatitis in severely obese children and adolescents undergoing sleeve gastrectomy. Surg Obes Relat Dis. 2017 Sep;13(9):1599-1609. doi: 10.1016/j.soard.2017.04.005. Epub 2017 Apr 7. PMID 28600116
- [Result] Alqahtani A, Elahmedi M, Qahtani AR. Laparoscopic Sleeve Gastrectomy in Children Younger Than 14 Years: Refuting the Concerns. Ann Surg. 2016 Feb;263(2):312-9. doi: 10.1097/SLA.0000000000001278. PMID 26496081
- [Result] Alqahtani AR, Elahmedi MO. Pediatric bariatric surgery: the clinical pathway. Obes Surg. 2015 May;25(5):910-21. doi: 10.1007/s11695-015-1586-x. PMID 25739495
- [Result] Alqahtani A, Alamri H, Elahmedi M, Mohammed R. Laparoscopic sleeve gastrectomy in adult and pediatric obese patients: a comparative study. Surg Endosc. 2012 Nov;26(11):3094-100. doi: 10.1007/s00464-012-2345-x. Epub 2012 May 31. PMID 22648112
- [Result] Alqahtani AR, Antonisamy B, Alamri H, Elahmedi M, Zimmerman VA. Laparoscopic sleeve gastrectomy in 108 obese children and adolescents aged 5 to 21 years. Ann Surg. 2012 Aug;256(2):266-73. doi: 10.1097/SLA.0b013e318251e92b. PMID 22504281
- [Result] Alqahtani AR, Elahmedi MO, Al Qahtani AR, Lee J, Butler MG. Laparoscopic sleeve gastrectomy in children and adolescents with Prader-Willi syndrome: a matched-control study. Surg Obes Relat Dis. 2016 Jan;12(1):100-10. doi: 10.1016/j.soard.2015.07.014. Epub 2015 Jul 22. PMID 26431633
- [Derived] Alqahtani AR, Elahmedi M, Abdurabu HY, Alqahtani S. Ten-Year Outcomes of Children and Adolescents Who Underwent Sleeve Gastrectomy: Weight Loss, Comorbidity Resolution, Adverse Events, and Growth Velocity. J Am Coll Surg. 2021 Dec;233(6):657-664. doi: 10.1016/j.jamcollsurg.2021.08.678. Epub 2021 Sep 23. PMID 34563670